CLINICAL TRIAL: NCT03554967
Title: Toluidine Blue Versus Frozen Sections for Assessment of Tumor Margins in Oral Squamous Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hana'a Hezam Ghaleb Algadi, principal investigator, Cairo University
Other Study IDs: 533
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Oral Squamous Cell Carcinoma
Keywords: Oral Squamous Cell Carcinoma; Toluidine Blue; Frozen Section; Tumor margin assessment
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to test the accuracy of toluidine blue in the assessment of intraoperative tumor margin after excision of oral squamous cell carcinoma(OSCC)in comparison to H&E stain on frozen section.

DETAILED DESCRIPTION:
The incidence of oral cancer remains high, it is ranked to be the sixth most common cancer worldwide, oral squamous cell carcinoma represent more than 90% of all oral malignances.

Standard treatment for oral squamous cell carcinoma is surgical resection with free margin. Negative margin status is an important for control local recurrence and improve outcome in squamous cell carcinoma of the head and neck. Hematoxylin and Eosin (H&E) Frozen section biopsy is useful tool for intraoperative assessment of resected margins and control of local recurrence, allowing for additional resection intraoperatively in case of positive margins. However in the least developed countries with limited resource, the frozen section is not available in a majority of centers, in addition to that if present in developed countries, it somewhat considered time and cost consumer.

Toluidine blue(TB) is metachromatic stain, easily available, economical, with high affinity for DNA and RNA. It is rapidly uptaken by malignant epithelium which contain quantitatively more nucleic acid than normal tissue. It has been widely used as screening tool for malignant and premalignant lesion.

The purpose of this study is to test the accuracy of toluidine blue in the assessment of intraoperative tumor margin after excision of oral squamous cell carcinoma(OSCC)in comparison to H&E stain on frozen section.

ELIGIBILITY:
Inclusion Criteria:

* Patient with biopsy-proven primary oral squamous cell carcinoma undergoing primary excision.

Exclusion Criteria:

* Patients with prior history of head and neck malignancy
* Patients with non-squamous cell carcinoma.
* Patients with previously undergone treatment (surgery and/or radio-/ chemotherapy) for the current oral squamous cell carcinoma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with biopsy-proven primary oral squamous cell carcinoma undergoing primary excision.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of toluidine blue VS frozen section for tumor margin assessment. | tumor margin will be assessed intraoperatively
  The diagnostic accuracy will be assessed by comparing the results of each technique with the final routine histopathological results.

CONTACTS AND LOCATIONS:
Overall Officials: Hana'a H Algadi, Msc student, Principal Investigator — Cairo University
Locations (1):
- Hana'a H Algadi, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Algadi HH, Abou-Bakr AA, Jamali OM, Fathy LM. Toluidine blue versus frozen section for assessment of mucosal tumor margins in oral squamous cell carcinoma. BMC Cancer. 2020 Nov 25;20(1):1147. doi: 10.1186/s12885-020-07644-0. PMID 33238944